CLINICAL TRIAL: NCT06050252
Title: A Phase II Trial of Durvalumab With Gemcitabine and Cisplatin as Neoadjuvant Therapy for High-Risk Resectable Intrahepatic Cholangiocarcinoma
Brief Title: Durvalumab With Gemcitabine and Cisplatin for the Treatment of High-Risk Resectable Liver Cancer Before Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-07031; NCI-2023-07031 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2024-0230; 10608 (Other: University of Texas MD Anderson Cancer Center LAO); 10608 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2023-09-21; First posted 2023-09-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Resectable Intrahepatic Cholangiocarcinoma
MeSH Terms: interventions — Biopsy; Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; durvalumab; Immunoglobulin G; Disulfides; Gemcitabine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (durvalumab, gemcitabine, cisplatin) (Experimental): Patients receive durvalumab IV over 60 minutes on day 1 with gemcitabine IV over 30 minutes and cisplatin IV over 60 minutes on days 1 and 8 for 4 cycles and then undergo surgical resection on study. Following surgery, patients may continue the durvalumab, gemcitabine and cisplatin regimen for up to 4 additional cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT scans and/or MRI scans and blood sample collection throughout study, as well as tissue biopsies during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Biological: Durvalumab; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Procedure: Resection

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Procedure: Magnetic Resonance Imaging — Undergo MRI scan
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection

SUMMARY:
This phase II trial tests how well giving durvalumab with standard chemotherapy, gemcitabine and cisplatin, before surgery works in treating patients with high risk liver cancer (cholangiocarcinoma) that can be removed by surgery (resectable). Durvalumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving durvalumab with gemcitabine and cisplatin before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed in patients with high risk resectable cholangiocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the proportion of patients who complete neoadjuvant therapy followed by curative intent surgical resection.

SECONDARY OBJECTIVES:

I. To determine the major pathologic response (MPR) rate. (Efficacy) II. To determine the proportion of patients who attain an R0 resection following neoadjuvant therapy. (Efficacy) III. To determine the radiological response rate after 2 and 4 cycles of neoadjuvant therapy. (Efficacy) IV. To determine the overall survival of patients receiving neoadjuvant therapy prior to curative intent surgical resection. (Efficacy) V. To determine the relapse free survival (RFS) of patients receiving neoadjuvant therapy prior to curative intent surgical resection. (Efficacy) VI. To estimate the incidence of adverse events during neoadjuvant therapy which would preclude completion of the neoadjuvant chemotherapy regiment as defined by grade 4 or above adverse events by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. (Feasibility) VII. To determine the proportion of patients who are able to start adjuvant therapy within 10 weeks of surgical resection. (Feasibility) VIII. To determine the proportion of patients who can complete 4 cycles of adjuvant therapy. (Feasibility) IX. To determine the efficacy of therapy in different molecular subtypes (by deoxyribonucleic acid [DNA] profiling, ribonucleic acid [RNA] profiling, and circulating tumor [ct]DNA-based minimal residual disease [MRD]). (Toxicity Profiles and Biomarkers) X. To compare pre- and post-neoadjuvant therapy changes in the phenotypic profiles of circulating immune cells. (Toxicity Profiles and Biomarkers) XI. To correlate ctDNA-based MRD, tissue and blood based immune biomarkers, and body composition with the primary/secondary endpoints. (Toxicity Profiles and Biomarkers)

EXPLORATORY OBJECTIVES:

I. Quantitative European Association for the Study of the Liver (qEASL)-based 3 dimensional (3D) enhancement measurement will be used as a surrogate marker of pathological response.

II. The primary and secondary outcomes will be associated with the visceral abdominal fat, subcutaneous abdominal fat, and muscle at the level of L2/L3.

OUTLINE:

Patients receive durvalumab intravenously (IV) over 60 minutes on day 1 with gemcitabine IV over 30 minutes and cisplatin IV over 60 minutes on days 1 and 8 for 4 cycles and then undergo surgical resection on study. Following surgery, patients may continue the durvalumab, gemcitabine and cisplatin regimen for up to 4 additional cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) scans and/or magnetic resonance imaging (MRI) scans and blood sample collection throughout study, as well as tissue biopsies during screening and on study.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 5 years and then yearly.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed intrahepatic cholangiocarcinoma (iCCA) that is resectable by imaging evaluation. Choice of staging modality is left up to the discretion of the treatment team; we favor high-quality CT scan of the chest/abdomen/pelvis with liver or biliary protocol. Eligibility will be confirmed through central imaging review.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 10 mm (>= 1 cm) with CT scan, MRI, or calipers by clinical exam.
* Patients must be an acceptable risk surgical candidate at the time of enrollment, as determined by a board-certified surgeon with expertise in hepatobiliary surgery.
* High-risk iCCA is defined as the presence of any of these factors:

  * Tumor size > 5 cm.
  * Multifocality or satellitosis limited to the same lobe.
  * Vascular invasion.
  * Suspected or confirmed (via biopsy) regional lymph node metastases.

    * Suspected is defined as lymph nodes that are deemed suspicious for metastasis based on large size (criteria vary per anatomical location; 6-10 mm for abdominal and 8-10 mm for pelvic), enhancement pattern, and shape. These may also include lymph nodes that display fludeoxyglucose F 18 (FDG)-avidity on positron emission tomography (PET) scan, if obtained, in the course of disease work-up (not mandatory).
  * CA 19-9 > 200 U/mL.
* Patients are treatment naïve for iCCA.
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of durvalumab (MEDI4736) in combination with cisplatin and gemcitabine in patients < 18 years of age, children are excluded from this study.
* Body weight > 30 kg.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%).
* Leukocytes >= 3,000/mcL.
* Hemoglobin >= 9.0 g/dL.
* Absolute neutrophil count >= 1,500/mcL.
* Platelets >= 100,000/mcL.
* Neuropathy grade =< 1 by CTCAE.
* Albumin >= 2.8 g/dL.
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) =< 3 × institutional ULN.
* Serum creatinine =< 1.5 x institutional ULN.
* Measured creatinine clearance > 60 mL/min or glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 (by the Cockcroft-Gault equation).
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Life expectancy >= 12 weeks.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. If non-protocol anticancer agents for non-study indications is required concurrently with the protocol therapy, the case should be discussed and approved by the study chair and the sponsor (Cancer Therapy Evaluation Program [CTEP]).
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Potential trial participants should have recovered from clinically significant adverse events of their most recent therapy/intervention prior to enrollment.
* Major surgical procedure (as defined by the Investigator) within 14 days prior to the first dose of durvalumab. Note: Local surgery of isolated lesions for palliative intent or biliary stents is acceptable.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection).
  * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent.
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab. Note: Patients, if enrolled, should not receive live vaccine whilst receiving durvalumab and up to 30 days after the last dose of durvalumab.
* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to durvalumab, gemcitabine, cisplatin, or other platinum-containing compounds.
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make this protocol unreasonably hazardous.
* Pregnant women are excluded from this study because durvalumab (MEDI4736) is an anti-PD-L1 monoclonal antibody agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with durvalumab, breastfeeding should be discontinued if the mother is treated with durvalumab. These potential risks may also apply to other agents used in this study. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after durvalumab administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of durvalumab.
* Patients with active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia.
  * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement.
  * Any chronic skin condition that does not require systemic therapy.
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
  * Patients with celiac disease controlled by diet alone.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* History of allogenic organ transplantation.
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-02-12 (Estimated); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who complete 4 cycles of neoadjuvant therapy followed by surgical resection | After surgical resection, up to week 18 after starting neoadjuvant therapy
  Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% confidence interval [CI]) will be reported. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.

SECONDARY OUTCOMES:
Major pathologic response (MPR) rate | After surgical resection, up to week 18 after starting neoadjuvant therapy
  MPR will be calculated based on the patients who can successfully undergo surgical resection. Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI) will be reported. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.
Proportion of patients who attain an R0 margin status after surgical resection | After surgical resection, up to week 18 after starting neoadjuvant therapy
  Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI) will be reported. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.
Radiological response rate | After 2 and 4 cycles of neoadjuvant therapy (cycle length=21 days)
  Defined as the percentage of patients with complete response, partial response, stable disease or progressive disease after neoadjuvant therapy by Response Evaluation Criteria in Solid Tumor (RECIST), modified RECIST and quantitative European Association for the Study of the Liver after completing 4 cycles of neoadjuvant therapy. Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI) will be reported. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.
Overall survival (OS) | From randomization to death, assessed up to 2 years
  OS, including treatment-related, and disease-related death will be assessed using immune RECIST. Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI) will be reported. Kaplan-Meier method will be used to estimate the survival curves. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.
Relapse free survival (RFS) | From surgery to recurrence of intrahepatic cholangiocarcinoma (iCCa), assessed up to 2 years
  Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% confidence interval (CI) will be reported. Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI) will be reported. Kaplan-Meier method will be used to estimate the survival curves. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.
Incidence of adverse events | Up to recurrence of iCCA
  Adverse events will be defined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI) will be reported. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.
Proportion of patients who are able to start adjuvant therapy | Up to 10 weeks after surgical resection
  Defined as the proportion of patients with Eastern Cooperative Oncology Group > 2, immunotherapy related adverse event > 3, any CTCAE > grade 3 that prevent from starting adjuvant therapy. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.
Proportion of patients who complete 4 cycles of adjuvant therapy | Up to week 12 after starting adjuvant therapy
  Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI will be reported. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.

OTHER OUTCOMES:
Tissue and blood based immune biomarkers | Up to week 12 after starting adjuvant therapy
  Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI) will be reported. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.
Tumor genomics, transcriptional profile and multiplex immunohistochemistry and multiplex immunofluorescence | Up to week 12 after starting adjuvant therapy
  Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI) will be reported. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.
Changes in circulating immune phenotypic profiles in the neoadjuvant phase | Up to week 12 after starting adjuvant therapy
  Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI) will be reported. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.
Circulating tumor deoxyribonucleic acid-based minimal residual disease correlated with pathological response and RFS | Up to week 12 after starting adjuvant therapy
  Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI) will be reported. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables.
Measures of body composition and fatty liver from imaging | Up to week 12 after starting adjuvant therapy
  Descriptive analysis will be used. Summary statistics (such as mean, median, range, proportion, as well as the associated 95% CI) will be reported. Regression models (such as the logistic regression for binary endpoints and the Cox regression for survival endpoints) will be constructed to assess the association between the primary/secondary endpoints and the prognostic or biomarker variables. Associate changes in subcutaneous abdominal fat, visceral abdominal fat, and muscle at the level of L3 with overall survival and recurrence free survival. Associate changes in body composition with toxicities that are observed during neoadjuvant therapy. Will calculate odds ratios here. Measure changes in the density of the liver before and after neoadjuvant therapy, and associate these with RECIST and responses radiographically. Will also associate density of the liver with pathological response to neoadjuvant therapy. Will use non-parametric statistical tests to do this (e.g., Wilcoxon).

CONTACTS AND LOCATIONS:
Overall Officials: Hop S Tran Cao, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (58):
- United States (58):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Los Angeles General Medical Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - NYP/Weill Cornell Medical Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm